CLINICAL TRIAL: NCT04028960
Title: Intranasal Insulin: A Novel Therapy for Hypoglycemia Unawareness in Type 1 Diabetes
Brief Title: IN Insulin in Type 1 Diabetes (T1D) Hypoglycemia Unawareness: Safety Only Phase
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding was rescinded
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A16-716
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-05

CONDITIONS: Type1diabetes
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): No active drug
  Interventions: Device: SipNose intranasal device
- Humulin-R (Experimental): Insulin
  Interventions: Drug: Regular insulin (Humulin-R), intranasal route; Device: SipNose intranasal device

INTERVENTIONS:
Drug: Regular insulin (Humulin-R), intranasal route — Humulin-R insulin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of diabetes.
  Arms: Humulin-R
Device: SipNose intranasal device — The SipNose device is an aerosol nasal delivery platform that uses pressurized delivery through the discharge of compressed air, resulting in an aerosol that delivers the drug in a narrow plume geometry, which targets the olfactory epithelium in the upper nasal cavity. From the olfactory epithelium, therapeutics rapidly reach the central nervous system, traveling extracellularly along the olfactory nerves. The device is not currently commercially available, but numerous studies have demonstrated its ability to intranasally deliver radiolabeled and therapeutic compounds to the brain.

SUMMARY:
The purpose of this study is to determine how Humulin-R regular insulin affects the body's ability to feel low blood sugar (hypoglycemia) when delivered intranasally compared to placebo in subjects with Type 1 Diabetes (T1D) with hypoglycemia awareness. The study will use continuous glucose monitoring (CGM) to collect this information. The study drug or placebo will be administered using an intranasal device.

DETAILED DESCRIPTION:
Hypoglycemia occurs with high frequency among patients with T1D. With repeated episodes of hypoglycemia, the counter-regulatory pathways to restore normal glucose are blunted, and patients can become unaware of the hypoglycemia. It is estimated that 40% of patients with T1D have hypoglycemia unawareness.

The study has the following objectives:

1. Primary:

   a. To assess non-inferiority of dangerous hypoglycemia with administration of intranasal insulin in T1D participants with intact awareness of hypoglycemia.
2. Secondary:

   1. To describe changes in overall glycemic control with administration of intranasal insulin in T1D participants with intact awareness of hypoglycemia
   2. To describe changes in hypoglycemia awareness with administration of intranasal insulin in T1D participants with intact awareness of hypoglycemia
   3. To describe changes in safety endpoints with administration of intranasal insulin in T1D participants with intact awareness of hypoglycemia.
3. Exploratory:

   1. To describe changes in memory, attention and executive function with administration of intranasal insulin in T1D participants with intact awareness of hypoglycemia

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18) with type 1 diabetes diagnosis and a duration of diabetes of at least 10 years
* Gold score <4
* HbA1c ≥6.5% within the last 3 months or at screen visit
* Stable insulin regimen (MDI or insulin pump) for at least 3 months, as deemed stable by principal investigator
* Depression/anxiety medications stable for at least 3 months
* Ability and willingness to wear CGM continuously during study participation
* Participants must use their own smartphone, and have the ability and willingness to use CGM smartphone applications compatible with their smartphone
* Ability and willingness to check self-monitoring of blood glucose (SMBG) using own supplies, as instructed by study staff
* Ability and willingness to document when having symptoms of hypoglycemia in the CGM smartphone app or in a diary
* Willing to operate insulin pump without threshold suspend feature or hybrid closed-loop, if applicable
* Proficient in speaking, reading and understanding English in order to complete surveys and testing of cognitive function
* Women of child-bearing age must agree to procure and use contraception throughout the study

Exclusion Criteria:

* Pregnancy or planning pregnancy
* eGFR ≤ 30 mL/min per 1.73 m2, if available from medical record
* Completed any other research study within 6 months of screening date
* Current or recent use within 3 months of an insulin delivery system that adjusts insulin in response to continuous glucose monitoring (CGM) data (such as an automated insulin delivery system like hybrid closed-loop insulin pump therapy)
* Known dementia or mild cognitive impairment diagnosis
* Diabetic ketoacidosis within the last 6 months
* Use of non-insulin medications to treat diabetes
* Those planning to change diet or exercise regimen during the study
* History of trans-sphenoidal surgery or surgery to the upper part of the nasal cavity, chronic sinusitis, severe deviated septum, or difficulty with smell and/or taste
* Severe psychiatric illness
* Allergy to adhesives, insulin or any components of insulin product
* Subject cannot adequately demonstrate ability to use and deploy the devices as determined by investigator
* Evidence of suicidality using the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Subject has history of any of the following: moderate to severe pulmonary disease, poorly controlled congestive heart failure, significant cardiovascular and/or cerebrovascular events within previous 6 months, condition known to affect absorption, distribution, metabolism, or excretion of drugs such as any hepatic, renal or gastrointestinal disease or any other clinically relevant abnormality or illness that inclusion would pose a safety risk to the subject as determined by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders L Carlson, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- Health Partners Institute dba International Diabetes Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Humulin-R Insulin: Participants first received a Placebo using the SipNose device twice daily for 14-20 days. After a washout period of 2 weeks, they received Humulin-R Insulin using the SipNose device twice daily for 14-20 days.
  SipNose intranasal device: The SipNose device is an aerosol nasal delivery platform that uses pressurized delivery through the discharge of compressed air, resulting in an aerosol that delivers the drug in a narrow plume geometry, which targets the olfactory epithelium in the upper nasal cavity. From the olfactory epithelium, therapeutics rapidly reach the central nervous system, traveling extracellularly along the olfactory nerves. The device is not currently commercially available, but numerous studies have demonstrated its ability to intranasally deliver radiolabeled and therapeutic compounds to the brain.
- Humulin-R Insulin, Then Placebo: Participants first received Humulin-R Insulin using the SipNose device twice daily for 14-20 days. After a washout period of 2 weeks, they received a Placebo using the SipNose device twice daily for 14-20 days.
  Regular insulin (Humulin-R), intranasal route: Humulin-R insulin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of diabetes.
  SipNose intranasal device: The SipNose device is an aerosol nasal delivery platform that uses pressurized delivery through the discharge of compressed air, resulting in an aerosol that delivers the drug in a narrow plume geometry, which targets the olfactory epithelium in the upper nasal cavity. From the olfactory epithelium, therapeutics rapidly reach the central nervous system, traveling extracellularly along the olfactory nerves. The device is not currently commercially available, but numerous studies have demonstrated its ability to intranasally deliver radiolabeled and therapeutic compounds to the brain.
Period: Overall Study
Arm/Group | Placebo, Then Humulin-R Insulin | Humulin-R Insulin, Then Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Four subjects were enrolled in the study. Two subjects started the study in the placebo arm and the other two started the study in the Humulin-R arm. During the study, each participant crossed over to the opposite arm of the study so that each subject participated in both arms of the study.
Groups:
- Humulin-R Insulin, Then Placebo: Participants first received Humilin-R Insulin using the SipNose device twice daily for 14-20 days. After a washout period of 2 weeks, they received a Placebo using the SipNose device twice daily for 14-20 days.
  Regular insulin (Humulin-R), intranasal route: Humulin-R insulin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of diabetes.
  SipNose intranasal device: The SipNose device is an aerosol nasal delivery platform that uses pressurized delivery through the discharge of compressed air, resulting in an aerosol that delivers the drug in a narrow plume geometry, which targets the olfactory epithelium in the upper nasal cavity. From the olfactory epithelium, therapeutics rapidly reach the central nervous system, traveling extracellularly along the olfactory nerves. The device is not currently commercially available, but numerous studies have demonstrated its ability to intranasally deliver radiolabeled and therapeutic compounds to the brain.
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Humulin-R Insulin | Humulin-R Insulin, Then Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (3.5) | 40.5 (6.4) | 52.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time With Dangerous Hypoglycemia
Description: Defined using percent time below range (<54 mg/dL), from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 0.57 (0.73) | 0.77 (1.08)

2. Secondary Outcome: Percent of Time With Blood Glucose 70-180 mg/dL
Description: Defined using percent of Blood Glucose 70-180 mg/dL from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 51.6 (16.3) | 49.5 (22.6)

3. Secondary Outcome: Percentage of Time With Blood Glucose <70 mg/dL
Description: Defined using percent of Blood Glucose <70 mg/dL from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 2.0 (1.7) | 1.6 (1.2)

4. Secondary Outcome: Percentage of Time Blood Glucose >180 mg/dL
Description: Percentage of time Blood Glucose >180 mg/dL from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 25.2 (2.1) | 26.3 (4.3)

5. Secondary Outcome: Percentage of Time With Blood Glucose >250 mg/dL
Description: Percentage of time with Blood Glucose >250 mg/dL from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 20.6 (17.7) | 21.9 (23.6)

6. Secondary Outcome: Percentage of Time Participant Had Active Sensor Wear
Description: Percentage of time Participant had Active Sensor Wear from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of time | 92.3 (9.2) | 93.5 (4.6)

7. Secondary Outcome: Mean Glucose From the Study Participants
Description: Mean Glucose from the Study Participants from real-time continuous glucose monitoring (CGM)
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
mg/dL | 188.4 (38.9) | 190.5 (50.9)

8. Secondary Outcome: Coefficient of Variation (%CV) of Blood Glucose Values From CGM Data
Description: The Coefficient of variation was calculated by dividing the standard deviation of blood glucose values by the mean of the blood glucose values based on data from the corresponding CGM readings.
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of CV
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of CV | 40.0 (6.5) | 37.8 (8.7)

9. Secondary Outcome: Glucose Management Indicator (GMI)
Description: An approximate HbA1c based upon real-time continuous glucose monitoring (CGM) values
Time Frame: Two 14-20 day treatment periods
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Placebo | Humulin-R
Number analyzed (Participants) | 4 | 4
percentage of HbA1c | 7.8 (0.9) | 7.9 (1.2)

ADVERSE EVENTS:
Time Frame: 5.5 months
Arm/Group | Placebo | Humulin-R
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Humulin-R (N=4)
Nose Bleeds (Skin and subcutaneous tissue disorders) | 3 (10) | 4 (7)
Nasal Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (7)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Respiratory/Sinus Symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The study team was unable to draw conclusions at this time regarding the cognitive testing performed due to abbreviated funding which led to a small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT04028960/Prot_SAP_000.pdf